CLINICAL TRIAL: NCT02403882
Title: An Analysis of Behavioral Economic Interventions at Client-Choice Food Pantries
Brief Title: Behavioral Economic Interventions at Food Pantries
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Auburn University (Other)
Collaborators: Cornell University (Other)
Responsible Party: Principal Investigator, Norbert L Wilson, Professor, Auburn University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AuburnU
Record Dates: First submitted 2015-03-18; First posted 2015-03-31 (Estimated); Last update posted 2016-04-26 (Estimated); Status verified 2016-04

CONDITIONS: Food Selection
Keywords: behavioral economics; food pantry; food choice
MeSH Terms: conditions — Food Preferences | interventions — Product Packaging; Costs and Cost Analysis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (5):
- Order (Experimental): The investigators arrange the placement of the targeted good to see if the order affects selection.
  Interventions: Behavioral: Order
- Packaging (Experimental): The investigators adjust the packaging of the targeted good to determine the effects on selection.
  Interventions: Behavioral: Packaging
- Pricing (Experimental): In food pantries, few products are priced. The investigators use pricing of products to determine its effect on selection.
  Interventions: Behavioral: Pricing
- Relative Proportions (Experimental): The investigators adjust the proportion of the products to determine the effect on the selection of the targeted product.
  Interventions: Behavioral: Relative Proportions
- Default Option (Experimental): The investigators provide a targeted product to subjects at one point. Later, investigators offer subjects the possibility to exchange the targeted product for a close substitute.
  Interventions: Behavioral: Default Option

INTERVENTIONS:
Behavioral: Order — In the order intervention, the investigators place the targeted product at the front of the line for the treatment. For the control, the investigators place the targeted product at the end of the line.
  Arms: Order
Behavioral: Packaging — In the packaging intervention, the investigator present the targeted product in the original package. In the control, the investigator repackage the targeted product in clear, plastic bags.
  Arms: Packaging
Behavioral: Pricing — In the pricing intervention, the investigators price all or targeted products in the treatment. In the control, the investigators do not price the products.
  Arms: Pricing
Behavioral: Relative Proportions — The investigators adjust the amount of the targeted good available relative to the other products. In the treatment, the targeted good is a larger proportion of the total goods offered in the section, while in the control the shares of the targeted and other goods are equal.
  Arms: Relative Proportions
Behavioral: Default Option — In an early site, the investigators offer a targeted product without an alternative. The subjects can accept or reject the offer. The subjects are told that an alternative product is available later. At the site where the alternative product is available, investigators offer subjects the opportunity to exchanged the targeted product for the alternative product.
  Arms: Default Option

SUMMARY:
The investigators run a series of behavioral economic interventions at client-choice food pantries to encourage clients to choose targeted foods.

DETAILED DESCRIPTION:
The study includes simple interventions at food pantries in New York State. In the initial phase, the investigators are testing the effect of order, packaging, pricing products, and relative proportion of products at a food pantry.

ELIGIBILITY:
Inclusion Criteria:

* Client in food pantry

Exclusion Criteria:

* Minors

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 443 (Estimated)
Dates: Start 2014-10; Primary Completion 2017-06 (Estimated); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
Number of Targeted Products Selected Relative to Others | up to 8 months
  As subjects choose products from sections of the food pantry, the investigators observe the selection of the targeted product among the other products available. If the targeted product is selected the investigators denote it with a one and zero otherwise. The investigators average the outcome over five and 10 subjects. The investigators also use probit and logistic models to estimate the probability of uptake.

CONTACTS AND LOCATIONS:
Overall Officials: Norbert L Wilson, PhD, Principal Investigator — Auburn University; David R. Just, PhD, Principal Investigator — Cornell University

REFERENCES:
- [Background] Wansink B, Just DR, Payne CR, Klinger MZ. Attractive names sustain increased vegetable intake in schools. Prev Med. 2012 Oct;55(4):330-332. doi: 10.1016/j.ypmed.2012.07.012. Epub 2012 Jul 27. PMID 22846502 (Retraction: PMID 29524989 Prev Med. 2018 May;110:116)
- [Background] Wansink B, Just DR, Payne CR. Can branding improve school lunches? Arch Pediatr Adolesc Med. 2012 Oct;166(10):1-2. doi: 10.1001/archpediatrics.2012.999. No abstract available. PMID 22911396 (Retraction: PMID 29053760 JAMA Pediatr. 2017 Dec 1;171(12 ):1230)
- [Background] Hanks AS, Just DR, Wansink B. Smarter lunchrooms can address new school lunchroom guidelines and childhood obesity. J Pediatr. 2013 Apr;162(4):867-9. doi: 10.1016/j.jpeds.2012.12.031. Epub 2013 Feb 22. PMID 23434267
- [Background] Wansink B, Just DR, Hanks AS, Smith LE. Pre-sliced fruit in school cafeterias: children's selection and intake. Am J Prev Med. 2013 May;44(5):477-80. doi: 10.1016/j.amepre.2013.02.003. PMID 23597811
- [Derived] Wilson NLW, Just DR, Swigert J, Wansink B. Food pantry selection solutions: a randomized controlled trial in client-choice food pantries to nudge clients to targeted foods. J Public Health (Oxf). 2017 Jun 1;39(2):366-372. doi: 10.1093/pubmed/fdw043. PMID 27173671